CLINICAL TRIAL: NCT04018859
Title: A Pilot Clinical Trial Investigating the Effect of Autologous Platelet-rich Plasma in Subjects With Mild to Moderate Eyebrow Hypotrichosis
Brief Title: Platelet-rich Plasma for Eyebrows
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00207701
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Eyebrow Hypotrichosis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Platelet-Rich Plasma (Experimental): Participants will receive intradermal injections of 2-3mL autologous PRP to eyebrows.Three treatments will be performed 1 month apart.
  Interventions: Device: Platelet Rich Plasma Prep System
- Placebo (sterile saline) (Placebo Comparator): Participants will receive intradermal injections of 2-3mL sterile saline to eyebrows.Three treatments will be performed 1 month apart.
  Interventions: Drug: Saline

INTERVENTIONS:
Device: Platelet Rich Plasma Prep System — intradermal injections of platelet rich plasma to the eyebrows
  Arms: Platelet-Rich Plasma
Drug: Saline — intradermal injections to the eyebrows
  Arms: Placebo (sterile saline)

SUMMARY:
The purpose of this study is to evaluate the effect of autologous platelet-rich plasma (PRP) in the treatment of mild to moderate eyebrow hypotrichosis.

This is a randomized clinical trial to evaluate the effect of autologous platelet rich plasma in subjects with mild to moderate eyebrow hypotrichosis. Approximately 40 subjects will be randomized to receive platelet-rich plasma (PRP) or saline injections. The study is designed as an 9-month study. This study was a pilot study designed to determine feasibility of this procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18-85 years old.
2. Subjects are in good health as judged by the investigator.
3. Patients with mild to moderate eyebrow hypotrichosis (modified GEyA grades of 3 and 4 at the time of screening, see Appendix A).
4. Those who have less eyebrows and therefore, desire to enhance eyebrows (modified GEyA grades of 3 and 4 at the time of screening, see Appendix A).
5. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator

Exclusion Criteria:

1. Patients with uncontrolled systemic disease (including alopecia areata or any other form of alopecia) which could inhibit hair growth
2. Patients with thrombocytopenia, platelet dysfunction, hypofibrinogenemia, anemia, cancer, active infections with Pseudomonas, Klebsiella, or Enterococcus, history of trichotillomania, thyroid diseases, eye diseases, atopic dermatitis, seborrheic dermatitis, lupus erythematosus, scleroderma, leprosy, or syphilis.
3. Patients who have started used agents that may affect eyebrow hair growth (e.g. minoxidil or bimatoprost) within 6 months of screening. Patients who have been using agents that may affect eyebrow hair growth for at least 12 months may be included if the patient agrees to continue their current dosing regimen for the duration of the study.
4. Known disease, infection, or abnormality in the treatment area or hair shaft
5. Patients with tattoos, scars, hyperpigmentation, or other features which could prevent accurate evaluation of hair growth in the eyebrow area.
6. Evidence of another skin condition affecting the treatment area that would interfere with clinical assessments
7. Unwilling to refrain from washing face or using face care products 24 hours before and after treatment visits
8. History of a clinically significant hematologic disorder as determined by the investigator.
9. Subjects currently receiving anticoagulant or anti-platelet therapy.
10. Subject is known to be HIV positive.
11. Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, etc.
12. Pregnant or breast feeding
13. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
14. Subjects who are unable to understand the protocol or give informed consent (including non-English speaking patients).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical change of eyebrow hypotrichosis, as determined by scoring photographs | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No